CLINICAL TRIAL: NCT01406145
Title: A Phase 1b, Multicenter, Double-Blind, Randomized, Placebo-Controlled, Sequential Dose Study of the Safety and Tolerability of ASP0777 in Subjects With Alzheimer's Disease on Donepezil
Brief Title: A Study of the Safety and Tolerability of ASP0777 in Subjects With Alzheimer's Disease (AD) Taking a Stable Dose of Donepezil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0777-CL-0030
Record Dates: First submitted 2011-07-06; First posted 2011-08-01 (Estimated); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Alzheimer's Disease
Keywords: ASP0777; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ASP0777 low dose (Experimental): ASP0777 low dose for 6 weeks
  Interventions: Drug: ASP0777
- ASP0777 low dose, then high dose (Experimental): ASP0777 low dose for 1 week and ASP0777 high dose for 5 weeks
  Interventions: Drug: ASP0777
- ASP0777 high dose (Experimental): ASP0777 high dose for 6 weeks
  Interventions: Drug: ASP0777
- Placebo (Placebo Comparator): Placebo for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP0777 — oral tablet
  Arms: ASP0777 high dose; ASP0777 low dose; ASP0777 low dose, then high dose
Drug: Placebo — oral tablet
  Arms: Placebo

SUMMARY:
This study is intended to determine the safety and tolerability of ASP0777 in subjects with Alzheimer's Disease (AD) taking a stable dose of donepezil.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a Mini-Mental Status Exam score of 18-26
* Subject has a diagnosis of "probable" Alzheimer's Disease
* Subject has used donepezil for at least 3 months and has been on a stable dose for at least 6 weeks prior to screening
* Subject has a reliable adult who is residing with him/her during the outpatient portion of the study
* Subject is medically stable
* Subject has adequate cognitive, hearing, vision, and language skills
* Subject is able to ingest oral tablets

Exclusion Criteria:

* Subject has received any investigational product in another clinical study or post-marketing clinical study within past 3 months
* Subject has any clinically significant abnormal laboratory tests
* Subject is a female who is pregnant, lactating or of childbearing potential who refuses to use a form of contraception during the study
* Subject has a history of a drug allergy or intolerance to memantine or a related compound
* Subject is currently using anti-dementia drugs (except for donepezil) or has used any such drugs within the last 4 weeks
* Subject has a score of 2 on item 16 of Cornell Scale for Depression in Dementia (CSDD) or has an overall CSDD score > 10
* Subject is using off-label medicines, non-medicinal compounds, or dietary aids/food supplements to improve cognition that have not been at a stable dose for at least 4 weeks prior to Screening and/or are anticipated to change dosing regimen during the study
* Subject has a history of drug or alcohol abuse within the past 12 months or subject consumes > 1 drink of alcohol daily, or is unable to refrain from alcohol during the study
* Subject is a current smoker or recently quit smoking (within the past 12 months)
* Subject has a clinically significant medical condition that is unstable or is likely to become unstable during the course of the study
* Subject has history of seizures, other than febrile seizures during infancy
* Subject has history of repeated falls within past 6 months
* Subject has a major psychiatric illness or has received treatment for symptoms of a major psychiatric illness within past 1 year. Mild psychiatric disorders are allowable

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06-16 (Actual); Primary Completion 2011-11-04 (Actual); Study Completion 2011-11-04 (Actual)

PRIMARY OUTCOMES:
Number and percentage of subjects with adverse events | Up to 56 Days

SECONDARY OUTCOMES:
Pharmacokinetic assessment of AUC, maximum concentration (Cmax), minimum concentration (Cmin) and time to maximum concentration (tmax) through analysis of blood samples | Up to 56 Days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (2):
- United States (2):
  - Pacific Research Network, Inc., San Diego, California
  - MD Clinical, Hallandale, Florida

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=296